CLINICAL TRIAL: NCT00083447
Title: A Phase III Multicenter Study of Intratumoral/Interstitial Therapy With TransMID™ Compared to Best Standard of Care in Patients With Progressive and/or Recurrent, Non-Resectable Glioblastoma Multiforme
Brief Title: Study of Therapy With TransMID™ Compared to Best Standard of Care in Patients With Glioblastoma Multiforme
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: This study has been withdrawn because the drug would not meet trial criteria for efficacy
Sponsor: Xenova Biomedix (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KSB311R/CIII/001; NCT00087230 (obsolete NCT alias)
Record Dates: First submitted 2004-05-24; First posted 2004-05-26 (Estimated); Last update posted 2009-01-07 (Estimated); Status verified 2008-01

CONDITIONS: Glioblastoma Multiforme
Keywords: brain tumor; GBM; glioblastoma; glioblastoma multiforme; brain cancer; treatment
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms | interventions — Tf-CRM107

INTERVENTIONS:
Drug: TransMID™

SUMMARY:
TransMID treatment or best standard of care for patients with advanced glioblastoma multiforme

Glioblastoma multiforme (GBM) is a type of brain tumour. GBM tumours are usually treated with surgery and radiotherapy. Unfortunately, this type of brain tumour may continue to grow or come back (recur) despite treatment.

This trial will compare a new drug called TransMID with the best standard treatment that is currently available. TransMID is a drug that is a combination of a protein called transferrin and a poison called diphtheria toxin.

Cancer cells need iron in order to continue to grow. They need more iron than normal cells. Transferrin helps cells to take up available iron. So the cancer cells are attached to the transferrin in TransMID, and the diphtheria poison kills them. The aim of this treatment is to kill the cancer cells while not affecting the normal brain cells. This treatment for brain tumours may have fewer side effects than other treatments because it targets cancer cells.

The best standard treatment will involve giving chemotherapy. You may have chemotherapy as part of the treatment when you are diagnosed. Or it may be kept in reserve to treat your brain tumour if it comes back or continues to grow. Your cancer specialist (consultant) will decide which chemotherapy drugs you should have.

DETAILED DESCRIPTION:
This is a Multicenter, open label, randomized study comparing TransMID™ with a chemotherapeutic regimen considered to be best standard of care and consisting of either nitrosoureas, platinum compounds, temozolomide, procarbazine, PCV, (procarbazine, lomustine (CCNU) & vincristine), CPT-11, or Etoposide. A planned interim analysis of the primary efficacy endpoint will be conducted after approximately 50% of the required events have been observed.

In order for a patient to be eligible for enrollment into this trial, he/she must be diagnosed with glioblastoma multiforme which has been confirmed histologically and have undergone conventional treatment, including surgery (biopsy or debulking) and/or radiation therapy and/or chemotherapy, have a recurrent and/or progressive tumor ≥1.0 cm and ≤4.0 cm in diameter.

ELIGIBILITY:
Inclusion Criteria:

1) Male or female at least 18 years of age 2) Histological results confirming GBM are available 3) Progressive GBM (≥ 25% increase in contrast enhanced tumor CSA compared to the nadir or smallest previous measured CSA) and/or recurrent GBM after conventional treatment, including surgery (biopsy or debulking surgery) and/or radiation therapy and/or chemotherapy 4) Pre-study MRIs used to determine current progression and/or recurrence of GBM are available to the Investigator and for independent confirmation of progression and/or recurrence 5) Patient is not considered a candidate for resection 6) If female of child-bearing potential, a reliable method of contraception must be combined with a negative pregnancy test before entering the study (female patients must be willing to use contraception for 2 months after the last treatment with TransMID™). Male patients must be willing to use a barrier method of contraception for up to 2 months after the last treatment with TransMID™ 7) Able and willing to follow instructions and comply with the protocol 8) Provide written informed consent prior to participation in the study 9) Karnofsky Performance Scale Score 70-100 10) Tumor characteristics: i) must be unifocal; and ii) must be unilateral and supratentorial; and iii) lesion must have a diameter (on contrast-enhanced MRI) ≥1.0 cm and ≤4.0 cm

Exclusion Criteria:

1) Anticipated life expectancy of less than 3 months 2 Infratentorial or intraventricular tumors 3) Presence of satellite tumors 4) Chemotherapy within 30 days prior to study entry or nitrosoureas or Mitomycin-C containing therapy within 42 days prior to study entry 5) External Beam irradiation within 60 days prior to study entry or stereotactic (gamma knife) radiosurgery within 90 days prior to study entry 6) Tumor surgery, tumor debulking or other neurosurgery within 5 days prior to study entry 7) Previous administration of TransMID™ 8) Previous enrollment in this study 9) Regional therapy including administration of biodegradable polymer wafers containing carmustine within 90 days prior to study entry or brachytherapy within 12 calendar months prior to study entry 10) Significant liver function impairment - AST or ALT > 2 times the upper limit of normal, total bilirubin > upper limit of normal 11) Hepatitis B surface antigen positive or positive Anti-Hepatitis C antibodies, or previous history of infectious Hepatitis (except previous Hepatitis A infection) 12) Significant renal impairment (serum creatinine > 1.7 mg/dL or 150 µmol/L) 13) Coagulopathy (prothrombin time [PT] or activated partial thromboplastin time [APTT] >1.5 times control) 14) Thrombocytopenia (platelet count < 100 x 103/μL or 100 x 109/L) 15) Granulocytopenia (absolute neutrophil count (ANC), < 1 x 103/μL or 1.0 x 109/L) 16) Severe acute infection 17) Medical condition that is considered an unacceptable anesthetic risk 18) Evidence of a mass effect on CT or MRI with more than a 5 mm midline shift and/or nausea, vomiting, reduced level of consciousness or clinically significant papilledema 19) Nursing or pregnant females. A pregnancy test will be performed on all females who are of child-bearing potential 20) Use of any investigational product and/or participation in another clinical research study within the last 30 days prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 323
Dates: Start 2004-05; Primary Completion 2006-03 (Actual); Study Completion 2007-06 (Estimated)

PRIMARY OUTCOMES:
Overall survival time i.e. to to death

SECONDARY OUTCOMES:
12 month survival rate
Tumor Response
Duration of Response
Time to Progression
6 and 12 month progression rates
Progression Free Survival
6 and 12 progression free survival rate
Quality of Life

CONTACTS AND LOCATIONS:
Locations (25):
- United States (24):
  - University of California-San Diego, La Jolla, California
  - University of Southern California, Los Angeles, California
  - University of Colorado Health Sciences Center, Denver, Colorado
  - Yale University, New Haven, Connecticut
  - Moffitt Cancer Center and Research Institute, Tampa, Florida
  - University of Chicago, Chicago, Illinois
  - University of Iowa Hospitals in Clinics, Cedar Rapids, Iowa
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Johns Hopkins Medical Center, Baltimore, Maryland
  - NINDS National Institutes of Health, Bethesda, Maryland
  - Fairview University Medical Center, Minneapolis, Minnesota
  - Saint Louis University Hospital, St Louis, Missouri
  - Cooper University Hospital, Camden, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Columbia University Medical Center, New York, New York
  - SUNY Upstate Medical University at Syracuse, Syracuse, New York
  - New York Medical College, Valhalla, New York
  - University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Legacy Emanuel Hospital and Technology Center, Portland, Oregon
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Semmes-Murphey Neurologic Institute, Memphis, Tennessee
  - University of Utah, Salt Lake City, Utah
  - Medical College of Virginia, Richmond, Virginia
- Neville Knuckey, MD, Nedlands, Western Australia, Australia